CLINICAL TRIAL: NCT06988202
Title: Comparative Effectiveness of Different Techniques for Repeat Ablation After Failed Initial Ablation for Persistent Atrial Fibrillation
Brief Title: Comparative Effectiveness of Different Techniques for Repeat Ablation of Atrial Fibrillation
Acronym: REPEAT-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan Steinberg, Research Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00010537
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; irregular heart beat; posterior wall isolation; pulmonary vein isolation; ablation; REPEAT-AF
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeat PVI without LA PWI (Other)
  Interventions: Procedure: Pulmonary Vein Isolation (PVI) without Left Atrial Posterior Wall Isolation (PWI)
- Repeat PVI with LA PWI (Other)
  Interventions: Procedure: Pulmonary Vein Isolation (PVI) with Left Atrial Posterior Wall Isolation (PWI)

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation (PVI) without Left Atrial Posterior Wall Isolation (PWI) — A doctor inserts a thin, flexible tube (called a catheter) through a blood vessel, usually in the groin, and guides it to the heart.
  Once the catheter is in place, the doctor uses pulsed field electroporation, heat (radiofrequency) or cold (cryoablation) to create small scars in the area where the pulmonary veins connect to the left atrium of the heart.
  These scars block the faulty electrical signals that cause AF, helping the heart maintain a normal rhythm.
  Arms: Repeat PVI without LA PWI
Procedure: Pulmonary Vein Isolation (PVI) with Left Atrial Posterior Wall Isolation (PWI) — PVI with an additional step where the doctor also isolates the back wall (posterior wall) of the left atrium.
  Arms: Repeat PVI with LA PWI

SUMMARY:
Atrial fibrillation (AF) is the most common type of irregular heartbeat doctors see. People with AF sometimes have a procedure called an ablation to help get their heart back into a normal rhythm. However, this treatment doesn't always work. This study is looking at whether adding an extra step to the usual ablation-specifically treating another area of the heart called the left atrial (LA) posterior wall-can help people feel better overall, compared to just repeating the standard pulmonary vein isolation ablation procedure.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years on date of consent
* One prior PVI ablation procedure > 3 months prior for persistent AF
* Recurrent paroxysmal or persistent symptomatic AF confirmed on ECG despite prior PVI
* Eligible for repeat ablation procedure
* Willingness to comply with all post-procedural follow-up requirements and to sign informed consent

Exclusion Criteria

* Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus)
* Prior ablation that included non-PVI LA ablation, or more than one prior PVI ablation procedure for persistent AF
* Prior surgical ablation for AF
* Contraindication to systematic anticoagulation
* LA diameter on echocardiogram > 6.0 cms
* LV ejection fraction < 35%
* NYHA class III-IV congestive heart failure
* Acute coronary syndrome or coronary artery bypass surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within 3 calendar months prior to consent date
* Enzyme-positive myocardial infarction within the past 3 calendar months prior to consent
* Severe aortic or mitral valvular heart disease eligible for percutaneous or surgical repair/replacement procedures
* Prior valve replacement with mechanical prosthesis
* Angiographic evidence of coronary disease that requires coronary revascularization and with likelihood of undergoing a CABG or PCI in the next 3 calendar months following consent date
* Stroke within 3 calendar months prior to consent date
* Any medical condition likely to limit survival to < 1 year
* Renal failure requiring dialysis at time of consent
* Pregnancy
* History of non-compliance to medical therapy
* Participation in other clinical trials (observational/lead registries are allowed) without approval from the CCRC
* Inability or unwillingness to provide informed consent
* Resides at such a distance from the enrolling site so travel to follow-up visits would be unusually difficult
* Does not anticipate residing in the vicinity of the enrolling site for the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change of Symptom Score on the Atrial Fibrillation Severity Scale (AFSS) | From Baseline to Month 12
  The AFSS is a 19-item self-report instrument measuring atrial fibrillation burden. It includes symptom severity (7 items), frequency/duration (4 items), health care utilization (4 items), and a global well-being visual analog scale. Items are summed into a composite total burden score, ranging from 0 to 100, with higher scores indicating greater symptom burden and healthcare impact.

SECONDARY OUTCOMES:
Time to First Atrial Fibrillation Episode Lasting > 30 Seconds | Up to 24 Months Following Randomization
  A proportion of patients that experience a first recurrence of atrial fibrillation or any atrial tachyarrhythmia lasting more than 30 seconds after repeat ablation (randomization), detected via monitoring.
Mean Total Atrial Fibrillation Burden from Serial Holter Recordings | From Randomization through Month 24
  Total cumulative duration (in minutes or hours) of atrial fibrillation or other atrial tachyarrhythmias recorded via serial Holter monitoring during the follow-up period.
Mean Total Number of Cardiovascular Health Care Utilization Events | From Randomization through Month 48
  Total number of cardiovascular-related hospital admissions, emergency room visits, and unplanned clinic visits, as recorded in medical records.
Mean Total Number of Major Clinical Events | From Randomization through Month 48
  The number of adjudicated major clinical events including decompensated heart failure requiring IV therapy, myocardial infarction, stroke/TIA, major bleeding, syncope, cardiac arrest, device implantation, repeat ablation, thromboembolic events, and serious procedural complications (e.g., atrio-esophageal fistula, tamponade).

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan Steinberg, MD, Principal Investigator — University of Rochester; Wojciech Zareba, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Clinical Cardiovascular Research Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided